CLINICAL TRIAL: NCT05274360
Title: Neuroscience-Based Aphasia Therapy Adapted to Remote, Mobile-Based Treatment
Brief Title: Remote Neurobased Approach to Aphasia Therapy
Acronym: RNAAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Bioengineering of Catalonia (Other)
Collaborators: Hospital Universitari Joan XXIII de Tarragona. (Other); Universitat Pompeu Fabra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RNAAT2021
Record Dates: First submitted 2021-11-16; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-12

CONDITIONS: Aphasia, Broca; Aphasia, Wernicke; Aphasia, Fluent; Aphasia, Nonfluent; Aphasia
MeSH Terms: conditions — Aphasia, Broca; Aphasia, Wernicke; Aphasia

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either an experimental group or a control group. In the experimental group the participants will receive mobile-based aphasia therapy for two weeks. In the control group participants will receive no additional therapy apart from the conventional aphasia therapy that they are already receiving.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Mobile evidence-based aphasia therapy
  Interventions: Behavioral: Mobile evidence-based aphasia therapy
- Control Group (Active Comparator): Conventional aphasia therapy
  Interventions: Behavioral: Conventional aphasia rehabilitation

INTERVENTIONS:
Behavioral: Mobile evidence-based aphasia therapy — Use of mobile application to practice language for 2 weeks with a recommendation of 2 sessions per day of 20 minutes. The Android application, which is a Unity-based 2D game, will be installed on the patient's own phone, and they will play individually with the support of a family member if needed. The patients are free to start and stop using the application at any time. The application is safe to use, and it consists of therapeutic training methods such as object-matching, word search, writing, and manual voice recordings.
  Arms: Experimental Group
Behavioral: Conventional aphasia rehabilitation — Control Group (conventional aphasia rehabilitation). No therapy as patients are in the chronic stage, where they do not receive healthcare rehabilitation training.
  Arms: Control Group

SUMMARY:
The purpose of this study is the development and validation of an evidence-based mobile application, based on the core premises of Intensive Language-Action Therapy (ILAT) for aphasia, for the training and improvement of chronic aphasia patients administered at the patient's home. It aims at testing the beneficial effect on the linguistic performance (as assessed by the Barcelona and CAL clinical tests) counteracting learned non-use and the usability of the application as a tool for training once discharged from hospital care.

DETAILED DESCRIPTION:
Acquired brain lesions such as stroke often result in the most common disabling neurological damages. Up to 42% of stroke patients suffer serious language deficits and patients are frequently left with chronic disabilities which adversely impact their quality of life. One of the main challenges in aphasia rehabilitation includes long-term effects. After a certain time (i.e., 3-6mo, chronic phase), the frequency of therapy will decrease or stop, even if the patient has not always reached the expected or desired level of recovery. After this, a body of evidence suggests that the person with aphasia might decrease the use of verbal language given the negative reinforcement when trying to use the deteriorated function and failing to achieve a successful communication. This might lead to relying on other forms of communication (e.g., gestures) and to a vicious cycle of deterioration of verbal skills known as Learned Non-Use principle. Together with the pandemic socioeconomic situation and limited resources at healthcare facilities, this calls for the need of effective and efficient interventions that can be deployed at the house of the patients, in the form of auto-administered therapy. Despite the limited exploration of portable technologies in aphasia recovery, their use has been extensive and successful in other domains such as motor rehabilitation. Importantly, patients with aphasia report that the number 1 topic they would like to know more about is how to keep recovering after therapy ends.

Following recent evidence on experience-dependent plasticity mechanisms for successful stroke recovery and well-established theory-grounded interventions, such as ILAT, the present study aims to study the usability and improvement potential of a mobile-based aphasia rehabilitation app for stroke patients, used at home. A previous collaboration between both centers (SPECS lab and Hospital Joan XIII) used a computer-based setup. In this study by Grechuta et al. (2019), the Rehabilitation Gaming System for aphasia (RGSa) shows positive significant results on language (P= 0.001) and communication (P<0.05) compared to conventional therapy in the long term (16 weeks). This study will assess the usability, risks, and clinical outcome of the same principles applied to a mobile application that is prescribed to be used at home for two twenty-minutes session per day during two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any type of aphasia
* 6 or more months have passed since the stroke (chronic stage)
* Age between 18 and 90 years

Exclusion Criteria:

* Non-compliance with some of the inclusion criteria
* Presence of major perceptual, cognitive, motor, cognitive or neuropsychological pathology that can interfere with aphasia or make it difficult to interact with the system, including severe forms of motor impairments and apraxia, visual processing deficits, planning deficits, learning deficits, memory deficits, or attentional deficits
* Inability to understand the study participation
* Patients with an Android phone or tablet

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Within-group changes of language function | This will be assessed one day before starting the treatment and at the end of the treatment protocol (after two weeks)
  Clinical scale for language (Barcelona Test) will be assessed at baseline T0 (prior to the use of the application) and T1 (after two weeks of use) for the experimental group.
  Scale from 0 (minimum) to 365 (maximum) where higher scores indicate a better outcome.
Within-group changes of communication | This will be assessed one day before starting the treatment and at the end of the treatment protocol (after two weeks)
  Clinical scale for communication (Communicative Activity Log; Pulvermüller et al., 2001b) will be assessed at baseline T0 (prior to the use of the application) and T1 (after two weeks of use) for the experimental group.
  Scale from 0 (minimum) to 5 (maximum) where higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Between-group change of language function | This will be assessed one day before starting the treatment and at the end of the treatment protocol (after two weeks)
  Clinical scale for language (Barcelona Test) will be assessed at baseline T0 (time 0) and T1 (time 1).
  Scale from 0 (minimum) to 365 (maximum) where higher scores indicate a better outcome.
Between-group change of communication | This will be assessed one day before starting the treatment and at the end of the treatment protocol (after two weeks)
  Clinical scale for communication (Communicative Activity Log; Pulvermüller et al., 2001b) will be assessed at baseline T0 (time 0) and T1 (time 1).
  Scale from 0 (minimum) to 5 (maximum) where higher scores indicate a better outcome.
Validation of usability of the technologies used | This will be assessed at the end of the treatment protocol (after two weeks) for the experimental group.
  System Usability Scale (SUS) will be used as a measure of usability of the application.
  Scale from 1 (minimum) to 5 (maximum) where higher scores indicate a better outcome.
Validation of usability, acceptability, and usefulness of the technologies used | This will be assessed at the end of the treatment protocol (after two weeks) for the experimental group.
  mHealth App Usability Questionnaire (MAUQ) (Zhou, Bao, Setiawan, Saptono, & Parmanto, 2019) will be used as a measure of usability, acceptability, and usefulness of the application.
  Scale from 1 (minimum) to 7 (maximum), where higher scores indicate a better outcome.
Amount and time of use | This will be measured continuously through the use of the application during the two weeks of use.
  Relationship between the total use of the application, measured in number of sessions and total time spent in minutes using the app, and improvement on the Barcelona test measured on scale from 0-365, where higher scores indicate a better outcome.
Cues used per practice session | This will be measured continuously through the use of the application during the two weeks of use.
  Count of cues used by the subjects during the primary sessions of use of the application and compared to the final sessions of use of the application.
Reaction time on tasks in the application | This will be measured continuously through the use of the application during the two weeks of use.
  Reaction time, measured in seconds, during the primary sessions of use of the application and compared to the final sessions of use of the application.
Subjects' own validation score of voice recordings | This will be measured continuously through the use of the application during the two weeks of use.
  The validation score recorded from the application during the primary sessions of use of the application and compared to the final sessions of use of the application. Measured between 0 and 1 and represents the subject's score of how well they performed the task and recording.
Risk assessment | This will be assessed at the end of the treatment protocol (after two weeks) for the experimental group.
  A custom questionnaire will be used to measure any risks associated with the use of the application.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Bioengineering of Catalonia - Specs Lab, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ameer K, Ali K. iPad Use in Stroke Neuro-Rehabilitation. Geriatrics (Basel). 2017 Jan 6;2(1):2. doi: 10.3390/geriatrics2010002. PMID 31011013
- [Background] Bakheit AM, Shaw S, Barrett L, Wood J, Carrington S, Griffiths S, Searle K, Koutsi F. A prospective, randomized, parallel group, controlled study of the effect of intensity of speech and language therapy on early recovery from poststroke aphasia. Clin Rehabil. 2007 Oct;21(10):885-94. doi: 10.1177/0269215507078486. PMID 17981847
- [Background] Brandenburg, C., & Power, E. (2019). Mobile Technology in Aphasia Rehabilitation: Current Trends and Lessons Learnt. Everyday Technologies in Healthcare, 293-317. https://doi.org/10.1201/9781351032186-16
- [Background] Engelter ST, Gostynski M, Papa S, Frei M, Born C, Ajdacic-Gross V, Gutzwiller F, Lyrer PA. Epidemiology of aphasia attributable to first ischemic stroke: incidence, severity, fluency, etiology, and thrombolysis. Stroke. 2006 Jun;37(6):1379-84. doi: 10.1161/01.STR.0000221815.64093.8c. Epub 2006 May 11. PMID 16690899
- [Background] Grechuta K, Rubio Ballester B, Espin Munne R, Usabiaga Bernal T, Molina Hervas B, Mohr B, Pulvermuller F, San Segundo R, Verschure P. Augmented Dyadic Therapy Boosts Recovery of Language Function in Patients With Nonfluent Aphasia. Stroke. 2019 May;50(5):1270-1274. doi: 10.1161/STROKEAHA.118.023729. PMID 30913976
- [Background] Grechuta K, Rubio Ballester B, Espin Munne R, Usabiaga Bernal T, Molina Hervas B, Mohr B, Pulvermuller F, San Segundo RM, Verschure PFMJ. Multisensory cueing facilitates naming in aphasia. J Neuroeng Rehabil. 2020 Sep 9;17(1):122. doi: 10.1186/s12984-020-00751-w. PMID 32907594
- [Background] Griffith, J. (2018). Encyclopedia of Clinical Neuropsychology. Encyclopedia of Clinical Neuropsychology, 2-4. https://doi.org/10.1007/978-3-319-56782-2
- [Background] Hallowell, B., & Chapey, R. (2012). Introduction to language intervention strategies in adult aphasia. Language Intervention Strategies in Aphasia and Related Neurogenic Communication Disorders: Fifth Edition, (November), 3-19.
- [Background] Hidaka Y, Han CE, Wolf SL, Winstein CJ, Schweighofer N. Use it and improve it or lose it: interactions between arm function and use in humans post-stroke. PLoS Comput Biol. 2012 Feb;8(2):e1002343. doi: 10.1371/journal.pcbi.1002343. Epub 2012 Feb 16. PMID 22761551
- [Background] Hilari K, Needle JJ, Harrison KL. What are the important factors in health-related quality of life for people with aphasia? A systematic review. Arch Phys Med Rehabil. 2012 Jan;93(1 Suppl):S86-95. doi: 10.1016/j.apmr.2011.05.028. Epub 2011 Nov 25. PMID 22119074
- [Background] Hinckley JJ, Hasselkus A, Ganzfried E. What people living with aphasia think about the availability of aphasia resources. Am J Speech Lang Pathol. 2013 May;22(2):S310-7. doi: 10.1044/1058-0360(2013/12-0090). PMID 23695907
- [Background] Hirsch T, Barthel M, Aarts P, Chen YA, Freivogel S, Johnson MJ, Jones TA, Jongsma MLA, Maier M, Punt D, Sterr A, Wolf SL, Heise KF. A First Step Toward the Operationalization of the Learned Non-Use Phenomenon: A Delphi Study. Neurorehabil Neural Repair. 2021 May;35(5):383-392. doi: 10.1177/1545968321999064. Epub 2021 Mar 11. PMID 33703971
- [Background] Holland A, Fromm D, Forbes M, MacWhinney B. Long-term Recovery in Stroke Accompanied by Aphasia: A Reconsideration. Aphasiology. 2017;31(2):152-165. doi: 10.1080/02687038.2016.1184221. Epub 2016 May 27. PMID 28713191
- [Background] Kim J, Thayabaranathan T, Donnan GA, Howard G, Howard VJ, Rothwell PM, Feigin V, Norrving B, Owolabi M, Pandian J, Liu L, Cadilhac DA, Thrift AG. Global Stroke Statistics 2019. Int J Stroke. 2020 Oct;15(8):819-838. doi: 10.1177/1747493020909545. Epub 2020 Mar 9. PMID 32146867
- [Background] Maceira-Elvira P, Popa T, Schmid AC, Hummel FC. Wearable technology in stroke rehabilitation: towards improved diagnosis and treatment of upper-limb motor impairment. J Neuroeng Rehabil. 2019 Nov 19;16(1):142. doi: 10.1186/s12984-019-0612-y. PMID 31744553
- [Background] Maier M, Ballester BR, Verschure PFMJ. Principles of Neurorehabilitation After Stroke Based on Motor Learning and Brain Plasticity Mechanisms. Front Syst Neurosci. 2019 Dec 17;13:74. doi: 10.3389/fnsys.2019.00074. eCollection 2019. PMID 31920570
- [Background] Mayo NE, Wood-Dauphinee S, Ahmed S, Gordon C, Higgins J, McEwen S, Salbach N. Disablement following stroke. Disabil Rehabil. 1999 May-Jun;21(5-6):258-68. doi: 10.1080/096382899297684. PMID 10381238
- [Background] Moffatt, K., Pourshahid, G., & Baecker, R. M. (2017). Augmentative and alternative communication devices for aphasia: the emerging role of "smart" mobile devices. Universal Access in the Information Society, 16(1), 115-128. https://doi.org/10.1007/s10209-015-0428-x
- [Background] Palmer R, Enderby P, Paterson G. Using computers to enable self-management of aphasia therapy exercises for word finding: the patient and carer perspective. Int J Lang Commun Disord. 2013 Sep-Oct;48(5):508-21. doi: 10.1111/1460-6984.12024. Epub 2013 Jun 18. PMID 24033650
- [Background] Pulvermuller F. Brain mechanisms linking language and action. Nat Rev Neurosci. 2005 Jul;6(7):576-82. doi: 10.1038/nrn1706. PMID 15959465
- [Background] Pulvermuller F, Berthier ML. Aphasia therapy on a neuroscience basis. Aphasiology. 2008 Jun;22(6):563-599. doi: 10.1080/02687030701612213. Epub 2008 May 21. PMID 18923644
- [Background] Pulvermuller F, Neininger B, Elbert T, Mohr B, Rockstroh B, Koebbel P, Taub E. Constraint-induced therapy of chronic aphasia after stroke. Stroke. 2001 Jul;32(7):1621-6. doi: 10.1161/01.str.32.7.1621. PMID 11441210
- [Background] Stahl B, Mohr B, Dreyer FR, Lucchese G, Pulvermuller F. Using language for social interaction: Communication mechanisms promote recovery from chronic non-fluent aphasia. Cortex. 2016 Dec;85:90-99. doi: 10.1016/j.cortex.2016.09.021. Epub 2016 Oct 15. PMID 27842269
- [Background] Tippett DC, Niparko JK, Hillis AE. Aphasia: Current Concepts in Theory and Practice. J Neurol Transl Neurosci. 2014 Jan;2(1):1042. PMID 24904925
- [Background] Vallila-Rohter S, Kiran S. Non-linguistic learning and aphasia: evidence from a paired associate and feedback-based task. Neuropsychologia. 2013 Jan;51(1):79-90. doi: 10.1016/j.neuropsychologia.2012.10.024. Epub 2012 Nov 2. PMID 23127795
- [Background] Zhou L, Bao J, Setiawan IMA, Saptono A, Parmanto B. The mHealth App Usability Questionnaire (MAUQ): Development and Validation Study. JMIR Mhealth Uhealth. 2019 Apr 11;7(4):e11500. doi: 10.2196/11500. PMID 30973342

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT05274360/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT05274360/ICF_001.pdf